CLINICAL TRIAL: NCT00147979
Title: Multicentric, Prospective, Randomized, Comparing Trial Between Bypass of the Femoropoplitea by PTFE and Heparin Bounded PTFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: JOTEC Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004/042
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PTFE with bounded heparin
  Interventions: Device: Bridging by PTFE with bounded heparin
- 2 (Active Comparator): PTFE without bounded heparin
  Interventions: Device: Bridging by PTFE without bounded heparin

INTERVENTIONS:
Device: Bridging by PTFE with bounded heparin — Bridging by PTFE with bounded heparin
  Arms: 1
Device: Bridging by PTFE without bounded heparin — Bridging by PTFE without bounded heparin
  Arms: 2

SUMMARY:
Comparison of two kinds of protheses for bridging of the femoropoplitea and/or femorotibiale: PTFE with or without bounded heparin

DETAILED DESCRIPTION:
Comparison of two kinds of protheses for bridging of the femoropoplitea and/or femorotibiale: PTFE with or without bounded heparin.

Evaluation of this comparison by clinical systems: ankle-arm index, duplex echo, follow-up of 2 years

ELIGIBILITY:
Inclusion Criteria:

* Patients with Peripheral Vascular Diseases with complaints of invalidating claudication, rest pain, ucera or gangrene
* Patients with damage of the arteria femoralis superficialis or poplitea, longer than 6 cm
* Reasonable outflow arteria
* Informed consent
* Patient able to take part in all follow-up examinations

Exclusion Criteria:

* Acute ischemia of the leg
* Patients with a ipsilateral inflow stenosis of more than 70% which can not be corrected before or during the surgery
* < 18 years
* Pregnancy
* Recent heart attack (< 1 month)
* Life expectancy less than 12 months
* Known allergy to heparin
* Known contrast allergy
* Known bleeding or coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2004-04; Primary Completion 2009-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Primary patency after 2 years | after 2 years

SECONDARY OUTCOMES:
Secondary patency | after 2 years
Limb salvage | after 2 years
Mortality | after 2 years
Re-intervention | after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vermassen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be